CLINICAL TRIAL: NCT06740929
Title: Hormonal Management of Heavy Menstrual Bleeding in Adolescents and Young Adults with and Without a Bleeding Disorder: a Prospective Observational Cohort Study
Brief Title: Hormonal Management of Heavy Menstrual Bleeding in Adolescents
Acronym: JAdoRE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Dehlia Moussaoui, Principal investigator, University Hospital, Geneva
Other Study IDs: 2024-01578
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Heavy Menstrual Bleeding; Bleeding Disorder
Keywords: heavy menstrual bleeding; bleeding disorder; adolescent; contraception; menstrual management
MeSH Terms: conditions — Menorrhagia; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thrombin generation markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to evaluate whether hormonal medications (such as contraceptive pill, patch, injectable progestins and hormonal intra-uterine device) have similar efficacy at managing heavy menstrual bleeding in adolescents with a bleeding disorder compared to those without. We also aim to assess the quality of life and hemoglobin and iron levels in this population.

DETAILED DESCRIPTION:
Adolescents with heavy menstrual bleeding and willing to start a hormonal medication to reduce menstrual flow are included. At baseline and during the study period, questionnaires and blood tests are performed. Adolescents with a bleeding disorder are compared to those without. Follow-up is 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults aged < 26yo
* Presenting to the gynecology consultation at HUG
* Diagnosed with heavy menstrual bleeding (PBAC > 100)
* Willing to initiate a hormonal medication to manage heavy menstrual bleeding

Exclusion Criteria:

* Pregnancy or planning to become pregnant during the study period
* Already using hormonal medication for menstrual management and/or contraception
* Known anatomical uterine pathology
* Using anticoagulant or antiaggregant agents

Max Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults presenting to the gynecology consultation at HUG.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of reduction in menstrual blood loss | 6 months after hormonal medication initiation
  Using PBAC (pictorial blood loss assessment chart)

SECONDARY OUTCOMES:
Percentage of reduction in menstrual blood loss | 3 months following hormonal medication initiation
  Using PBAC
Percentage of reduction in menstrual blood loss | 12 months after hormonal medication initiation
  Using PBAC
Quality of life | at baseline, 3 months, 6 months and 12 months
  QoL (measured by the Pediatric Quality of Life Inventory (PedsQL) for adolescents (13-18 years old) or young adults (19-25 years old)) ; range 0-100 with higher scores representing better quality of life.
Hemoglobin and ferritin levels changes | at baseline, 6 months and 12 months
  Blood samples to measure hemoglobin and ferritin
Changes in thrombin generation markers | at baseline and 6 months
  Blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided